CLINICAL TRIAL: NCT05061472
Title: The Influence of Combined Oral Contraceptives on Weight, Body Composition, Eating Behaviors, and Appetite in Pre-menopausal Women With Overweight or Obesity
Brief Title: A 6-month Observational Study on Combined Oral Contraceptives and Body Weight in Pre-Menopausal Women With Overweight or Obesity
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3969
Record Dates: First submitted 2021-09-16; First posted 2021-09-29 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Contraceptive Usage; Overweight or Obesity; Body Weight Changes; Appetitive Behavior; Eating Behavior
Keywords: Combined Oral Contraceptive Pill; Body Weight; Body Composition; Eating Behaviors; Appetite; Pre-menopausal Women; Overweight; Obesity; Non-Hormonal Contraception
MeSH Terms: conditions — Contraception Behavior; Overweight; Obesity; Body Weight Changes; Appetitive Behavior; Feeding Behavior; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined Oral Contraceptives: Pre-menopausal women with overweight or obesity who are newly initiating the combined oral contraceptive pill, Sprintec (norgestimate/ethinyl estradiol 0.25mg/35mcg)
- Nonhormonal Contraceptives (Control): Pre-menopausal women with overweight or obesity who are using non-hormonal methods of birth control

SUMMARY:
Approximately 15 million women of reproductive age women in the United States have overweight or obesity and use the combined estrogen and progestin oral contraceptive pill (COC). Although many women report weight gain as a side effect of COCs, a conclusive link between COC use and weight gain has not been established. This investigation will address a major gap in the literature by prospectively evaluating the influence of initiating a COC versus non-hormonal contraceptives (NHCs) on weight, body composition, eating behaviors, and appetite in pre-menopausal women with overweight or obesity. Aim 1 will assess the feasibility of recruiting and retaining a racially/ethnically diverse group of women with overweight and obesity while Aim 2 will explore changes in body weight, body composition, and cardiometabolic risks in these women; Aim 3 will explore changes in dietary and macronutrient energy intake, eating behaviors, and appetite in this subset of women. This research will help the investigators understand the extent to which COCs are associated with weight gain and help guide medical providers in counseling women with overweight and obesity on appropriate contraceptive methods.

DETAILED DESCRIPTION:
The overall objective of this feasibility pilot study is to prospectively evaluate the effects of initiating a combined estrogen and progestin oral contraceptive (COC) compared to a non-hormonal contraceptive (NHC) on body weight, body composition, eating behaviors, and appetite in pre-menopausal women with overweight or obesity. Nearly half of the 61 million U.S. women of reproductive age have overweight or obesity, placing them and their offspring at an elevated lifetime risk of adverse cardiometabolic and health outcomes. Notably, ~15-20% of reproductive-aged women use COCs. Though many women anecdotally report weight gain as a side effect of COCs, a conclusive link between COC use and weight gain has not been established. Previous studies evaluating COCs and weight change have excluded women with obesity, who may be at greater risk for contraceptive-associated weight gain. Given the widespread use of COCs, it is critical to understand the extent to which these contraceptive methods may be associated with weight gain and correlated cardiometabolic health risks in reproductive age women with established overweight or obesity.

The reproductive hormonal profile of COC users differs substantially from that of normally cycling women. A recent study of seven typical COCs found that while median exposure to synthetic estrogens across a 28-day cycle was similar to median endogenous estrogen exposure, median synthetic progestin exposure was 4-fold higher than median endogenous progesterone exposure. COCs also lead to daily spikes in serum estrogen and progestin levels, unlike the gradual increase and cyclic patterns of endogenous hormones that characterize a normal menstrual cycle. COCs may impact weight via changes in appetite and satiety due to supraphysiologic systemic levels of reproductive hormones. For example, progesterone has been shown to increase appetite and trigger binge- or emotional-eating. The principal investigator has reported that use of COCs was associated with greater weight regain over 1 year after weight loss in women with overweight and obesity enrolled in a behavioral weight loss program. However, no studies have prospectively evaluated changes in body weight, cardiometabolic risk factors, and eating behaviors in women with overweight or obesity initiating COC vs. those using NHCs.

This study's overall hypothesis is that initiation of COCs in women with overweight or obesity will be associated with greater weight gain and increases in cardiometabolic health risks than use of NHCs over 6 months. The investigators will recruit pre-menopausal women with overweight or obesity who have already elected to initiate COCs as well as a control group of age and BMI matched NHC users. The investigators will evaluate the feasibility of recruiting women initiating a COC and women using NHCs into a prospective, observational study as well as the feasibility of evaluating changes in weight, body composition, eating behaviors, and appetite over 6 months from COC initiation. The investigators propose the following specific aims:

Aim 1: Assess the feasibility of recruiting and retaining a racially/ethnically diverse group of pre-menopausal women with overweight or obesity initiating COCs compared to age- and BMI-matched NHC users. The investigators aim to recruit ~10 women per month for 6 months (N=24; n=12 COCs, n=12 NHCs; >20% in each group of African American or Hispanic race/ethnicity) and assess feasibility of completion of outcome measures. The investigators hypothesize that at least 80% of participants will continue their chosen contraceptive method and complete outcome measures within a 2-week window at 6 months.

Exploratory Aim 2: Explore the influence of COC vs. NHC use on body weight, body composition, and cardiometabolic risk factors. The investigators hypothesize that women with overweight or obesity initiating COCs will exhibit greater increases in body weight, fat mass, homeostatic model assessment for insulin resistance (HOMA-IR), triglycerides, and blood pressure compared to age- and BMI-matched NHC users.

Exploratory Aim 3: Explore the influence of COC vs. NHC use on energy intake (EI), eating behaviors, and appetite. The investigators hypothesize that women with overweight or obesity initiating COCs will have greater increases in dietary energy and fat/carbohydrate intake, hunger, disinhibition, reward-based eating, emotional eating, binge eating, and food cravings at 6 months compared to age- and BMI-matched NHC users.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 18-40 years
* Overweight or class I-III obesity (BMI 25-45 kg/m2)
* Free of major psychiatric illnesses
* Electing to start the Sprintec (norgestimate/ethinyl estradiol 0.25mg/35mcg) COC
* Using non-hormonal forms of contraception: copper intrauterine device (Paragard), male condoms, tubal ligation, partner vasectomy, withdrawal/natural family planning, spermicide, abstinence, or other NHCs as determined by the investigators

Exclusion Criteria:

* Diabetes
* Use of medications thought to affect body weight, energy intake, glycemic parameters, or estrogen (i.e. systemic glucocorticoids, stimulants, weight loss pharmacotherapy, metformin)
* History of weight loss surgery
* History of polycystic ovarian syndrome
* History of congenital adrenal hyperplasia
* Use of a different COC or hormonal contraception method within the past 3 months
* Planning pregnancy
* Planning to stop contraceptive within the next 6 months
* Planning to change diet or join a weight loss program or research study within the next 6 months
* Recent therapeutic abortion or miscarriage in the past 1 month if fetal gestational age <10 weeks, or 3 months if fetal gestational age >10 weeks
* Pregnancy with delivery in the past 6 months
* Currently lactating
* People with pregnancy potential who were assigned female at birth and either currently using or planning to use gender-affirming hormone therapy in the next 6 months
* Use of other forms of reproductive hormones such as testosterone or dehydroepiandrosterone (DHEA)
* Current tobacco use

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The study will be performed in a cohort of up to 64 females of reproductive age, age 18-40 years, with overweight or class I-III obesity (BMI 25-45 kg/m2) who initiate the Sprintec COC pill or remain on a NHC
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnin Zaman, MD, Principal Investigator — University of Colorado, Denver; Victoria A Catenacci, MD, Study Chair — University of Colorado, Denver; Elizabeth A Thomas, MD, Study Chair — University of Colorado, Denver; Aaron Lazorwitz, MD, Study Chair — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Comprehensive Women's Health Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Cedergren MI. Maternal morbid obesity and the risk of adverse pregnancy outcome. Obstet Gynecol. 2004 Feb;103(2):219-24. doi: 10.1097/01.AOG.0000107291.46159.00. PMID 14754687
- [Background] Sebire NJ, Jolly M, Harris JP, Wadsworth J, Joffe M, Beard RW, Regan L, Robinson S. Maternal obesity and pregnancy outcome: a study of 287,213 pregnancies in London. Int J Obes Relat Metab Disord. 2001 Aug;25(8):1175-82. doi: 10.1038/sj.ijo.0801670. PMID 11477502
- [Background] Koliaki C, Liatis S, Kokkinos A. Obesity and cardiovascular disease: revisiting an old relationship. Metabolism. 2019 Mar;92:98-107. doi: 10.1016/j.metabol.2018.10.011. Epub 2018 Nov 3. PMID 30399375
- [Background] Coney P, Washenik K, Langley RG, DiGiovanna JJ, Harrison DD. Weight change and adverse event incidence with a low-dose oral contraceptive: two randomized, placebo-controlled trials. Contraception. 2001 Jun;63(6):297-302. doi: 10.1016/s0010-7824(01)00208-6. PMID 11672550
- [Background] Gallo MF, Lopez LM, Grimes DA, Carayon F, Schulz KF, Helmerhorst FM. Combination contraceptives: effects on weight. Cochrane Database Syst Rev. 2014 Jan 29;2014(1):CD003987. doi: 10.1002/14651858.CD003987.pub5. PMID 24477630
- [Background] Moore LL, Valuck R, McDougall C, Fink W. A comparative study of one-year weight gain among users of medroxyprogesterone acetate, levonorgestrel implants, and oral contraceptives. Contraception. 1995 Oct;52(4):215-9. doi: 10.1016/0010-7824(95)00189-h. PMID 8605778
- [Background] Redmond G, Godwin AJ, Olson W, Lippman JS. Use of placebo controls in an oral contraceptive trial: methodological issues and adverse event incidence. Contraception. 1999 Aug;60(2):81-5. doi: 10.1016/s0010-7824(99)00069-4. PMID 10592854
- [Background] Risser WL, Gefter LR, Barratt MS, Risser JM. Weight change in adolescents who used hormonal contraception. J Adolesc Health. 1999 Jun;24(6):433-6. doi: 10.1016/s1054-139x(98)00151-7. PMID 10401972
- [Background] Mayeda ER, Torgal AH, Westhoff CL. Weight and body composition changes during oral contraceptive use in obese and normal weight women. J Womens Health (Larchmt). 2014 Jan;23(1):38-43. doi: 10.1089/jwh.2012.4241. Epub 2013 Oct 24. PMID 24156617
- [Background] Gallo MF, Grimes DA, Schulz KF, Helmerhorst FM. Combination estrogen-progestin contraceptives and body weight: systematic review of randomized controlled trials. Obstet Gynecol. 2004 Feb;103(2):359-73. doi: 10.1097/01.AOG.0000107298.29343.6a. PMID 14754709
- [Background] Grandi G, Piacenti I, Volpe A, Cagnacci A. Modification of body composition and metabolism during oral contraceptives containing non-androgenic progestins in association with estradiol or ethinyl estradiol. Gynecol Endocrinol. 2014 Sep;30(9):676-80. doi: 10.3109/09513590.2014.922947. Epub 2014 Jun 11. PMID 24918262
- [Background] Lovett JL, Chima MA, Wexler JK, Arslanian KJ, Friedman AB, Yousif CB, Strassmann BI. Oral contraceptives cause evolutionarily novel increases in hormone exposure: A risk factor for breast cancer. Evol Med Public Health. 2017 Jun 5;2017(1):97-108. doi: 10.1093/emph/eox009. eCollection 2017. PMID 28685096
- [Background] Fleischman DS, Navarrete CD, Fessler DM. Oral contraceptives suppress ovarian hormone production. Psychol Sci. 2010 May;21(5):750-2; author reply 753. doi: 10.1177/0956797610368062. Epub 2010 Apr 22. No abstract available. PMID 20483856
- [Background] Leeners B, Geary N, Tobler PN, Asarian L. Ovarian hormones and obesity. Hum Reprod Update. 2017 May 1;23(3):300-321. doi: 10.1093/humupd/dmw045. PMID 28333235
- [Background] Caldwell AE, Zaman A, Ostendorf DM, Pan Z, Swanson BB, Phelan S, Wyatt HR, Bessesen DH, Melanson EL, Catenacci VA. Impact of Combined Hormonal Contraceptive Use on Weight Loss: A Secondary Analysis of a Behavioral Weight-Loss Trial. Obesity (Silver Spring). 2020 Jun;28(6):1040-1049. doi: 10.1002/oby.22787. PMID 32441474
- See also: Current Contraceptive Status Among Women Aged 15-49: United States, 2015-2017 — https://www.cdc.gov/nchs/data/databriefs/db327-h.pdf
- See also: Contraceptive Use in the United States by Demographics — https://www.guttmacher.org/fact-sheet/contraceptive-use-united-states

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Oral Contraceptives: Pre-menopausal women with overweight or obesity who are newly initiating the norgestimate/ethinyl estradiol 0.25mg/35mcg combined oral contraceptive pill.
Period: Month 0 (Baseline)
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Month 3
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Started | 10 | 10
Completed (One participant completed 3-month measures and then withdrew due to worsening mental health after completion of outcome measures at this timepoint.) | 10 | 10
Not Completed | 0 | 0
Period: Month 6 (Final)
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.4) | 30.5 (4.0) | 29.9 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Highest Level of School Completed [Count of Participants; unit: Participants]
  12th Grade | 1 | 0 | 1
  2-year College | 1 | 0 | 1
  4-year College | 4 | 5 | 9
  Master's Degree | 2 | 5 | 7
  Doctorate Degree | 1 | 0 | 1
  Other | 1 | 0 | 1
Annual Household Income [Count of Participants; unit: Participants]
  < $25,000 | 1 | 0 | 1
  $25,000-$45,000 | 0 | 0 | 0
  $45,001-$70,000 | 6 | 5 | 11
  $70,001-$110,000 | 1 | 4 | 5
  > $100,001 | 2 | 1 | 3
Marital Status [Count of Participants; unit: Participants]
  Single | 3 | 5 | 8
  Committed Relationship | 5 | 3 | 8
  Married | 2 | 2 | 4
  Separated | 0 | 0 | 0
Reported overweight as child? [Count of Participants; unit: Participants]
  Yes | 7 | 6 | 13
  No | 3 | 4 | 7
Highest reported non-pregnant adult weight [Median (Inter-Quartile Range); unit: pounds] | 185 [185 to 200] | 193 [175 to 205] | 188 [181 to 205]
Age at menarche [Median (Inter-Quartile Range); unit: years] | 11.5 [11 to 13] | 12 [10 to 13] | 12 [11 to 13]
Normal periods in the last year? [Count of Participants; unit: Participants]
  Yes | 8 | 8 | 16
  No | 2 | 2 | 4
Ever pregnant? [Count of Participants; unit: Participants]
  Yes | 3 | 0 | 3
  No | 7 | 10 | 17
Currently Exercising? [Count of Participants; unit: Participants]
  Yes | 6 | 9 | 15
  No | 4 | 1 | 5
Currently Using... [Number; unit: participants]
  Tobacco | 0 | 0 | 0
  Alcohol | 9 | 8 | 17
  Recreational Drugs | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Premenopausal Women With Overweight/Obesity Who Initiated a COC vs. Continued NHC Use, Enrolled and Remained in This Study, and Completed Outcome Measures
Description: The investigators aim to recruit ~10 women per month for 6 months (N=24; n=12 COCs, n=12 NHCs; >20% in each group of African American or Hispanic race/ethnicity) and assess feasibility of completion of outcome measures. The investigators hypothesize that at least 80% of participants will continue their chosen contraceptive method and complete outcome measures within a 2-week window at 6 months.
  The 6-month date was calculated as baseline outcome date + 182 days. A 2-week window was considered a +/- 14 days from the calculated 6-month outcome date.
Time Frame: Baseline, Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Number analyzed (Participants) | 10 | 10
Participants
  Completed 6 Month Measures within a 2-week Time Frame from Baseline Outcome Measure Date | 9 | 10
  Did Not Complete 6-Month Measures within a 2-week Time Frame from Baseline Outcome Measure Date | 1 | 0

2. Other Pre Specified Outcome: Body Weight
Description: Body Weight in pounds (lbs)
Time Frame: 6 Months
Measure: Median (90% Confidence Interval); unit: pounds
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Number analyzed (Participants) | 10 | 10
pounds
  Month 0 | 186.3 [175.8 to 194.2] | 185.1 [163.3 to 198.5]
  Month 6 | 182.5 [180.9 to 184.6] | 187.7 [167.3 to 198.9]

3. Other Pre Specified Outcome: BMI
Description: Body Mass Index (BMI [kg/m^2]) from dual x-ray absorptiometry
Time Frame: 6 Months
Measure: Median (90% Confidence Interval); unit: kg/m^2
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Number analyzed (Participants) | 10 | 10
kg/m^2
  Month 0 | 30.1 [28.9 to 33.0] | 30.5 [28.6 to 31.1]
  Month 6 | 29.3 [28.6 to 31.1] | 30.8 [28.8 to 33.4]

4. Other Pre Specified Outcome: Percent Body Fat
Description: % Body Fat (Fat Mass/Total Mass) as assessed on dual x-ray absorptiometry (DXA)
Time Frame: 6 Months
Measure: Median (90% Confidence Interval); unit: percent
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
Number analyzed (Participants) | 10 | 10
percent
  Month 0 | 42.5 [41.1 to 43.8] | 41.3 [38.4 to 44.6]
  Month 6 | 44.4 [41.0 to 45.1] | 43.1 [40.7 to 44.9]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Combined Oral Contraceptives | Nonhormonal Contraceptives (Control)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Oral Contraceptives (N=10) | Nonhormonal Contraceptives (Control) (N=10)
Changes in Mental Health (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT05061472/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT05061472/ICF_001.pdf